CLINICAL TRIAL: NCT05591092
Title: Radioiodine Scanning for Pre-Surgical Evaluation of Follicular Thyroid Nodules
Brief Title: Radioiodine Planar and a SPECT/CT Imaging With Iodine-123 for Evaluation of Follicular Thyroid Nodules Prior to Surgery
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 20-010663; NCI-2022-03573 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-10-18; First posted 2022-10-24 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Thyroid Gland Follicular Carcinoma
MeSH Terms: conditions — Adenocarcinoma, Follicular | interventions — Iodine-123; X-Rays; Photons

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (I-123, planar imaging, SPECT/CT scan): Patients receive iodine-123 PO and then undergo planar imaging and a SPECT/CT scan on study.
  Interventions: Procedure: Computed Tomography; Radiation: Iodine I-123; Procedure: Planar Imaging; Procedure: Single Photon Emission Computed Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo a SPECT/CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Radiation: Iodine I-123 — Given PO
  Other Names: I-123; Iodine 123; Iodine I 123; Isotope of Mass 123
Procedure: Planar Imaging — Undergo planar imaging
Procedure: Single Photon Emission Computed Tomography — Undergo a SPECT/CT scan
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon

SUMMARY:
This study evaluates radioiodine planar and SPECT/CT imaging with iodine-123 in patients with follicular thyroid nodules prior to surgery. Because biopsy alone is not sufficient to distinguish between malignant follicular thyroid nodules and benign follicular thyroid nodules, patients with follicular thyroid lesions are referred for surgery for further evaluation. A non-invasive imaging method that can accurately determine malignancy in follicular thyroid nodules would be valuable in patient management and could potentially spare patients unnecessary surgery. Planar imagine uses a gamma camera to obtain 2D images and SPECT/CT imaging is a special type of CT scan in which a small amount of a radioactive drug is injected into a vein and a scanner is used to make detailed images of areas inside the body where the radioactive material is taken up by the tumor cells. Radioiodine planar and SPECT/CT imaging may be more accurate in distinguishing between benign follicular thyroid nodules and malignant follicular thyroid nodules to help reduce the need for surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the proportion of benign nodules appearing as hot/warm on radioiodine scans (nodule uptake >= uptake in normal thyroid tissues).

II. To identify a possible relationship between iodine-123 (I-123) uptake on planar and single-photon emission computerized tomography (SPECT)/computerized tomography (CT) images and malignancy on surgical pathology in thyroid nodules that were previously identified by fine-needle aspiration (FNA) as indeterminate follicular neoplasm.

III. Examine correlations between intensity of uptake in follicular nodules before surgery (standard uptake values [SUV] on the quantitative reconstructions from our Veriton SPECT/CT scanner and nodule-to-normal thyroid background ratios on planar and SPECT images) and pathology findings and determine a SUV threshold that best distinguishes between benign and malignant nodules.

IV. Compare the usefulness of conventional planar imaging versus SPECT/CT imaging for thyroid nodules, in order to inform our optimal clinical protocol.

V. Establish an imaging protocol best suited for measuring uptake in small thyroid nodules.

OUTLINE:

Patients receive iodine-123 orally (PO) and then undergo planar imaging and a SPECT/CT scan on study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Any gender
* Patients will have had no therapy for their thyroid nodule prior to enrollment
* Negative urine pregnancy test within 48 hours before the administration of radiopharmaceutical in women of childbearing potential
* Follicular neoplasm or suspicious of follicular neoplasm, cytopathology on biopsy of thyroid nodule
* Any outside fine needle aspiration (FNA) reports are to be reviewed by a Mayo pathologist
* Nodules 1-4 cm with solid appearance on ultrasound
* Ultrasound images and report documented in medical record, including the size of the nodule and location (upper, mid or lower portion of the thyroid lobe)
* At least 2/3 of either thyroid lobe without nodules should be present to allow for the measurement of uptake in unaffected thyroid tissue
* Thyroid stimulating hormone (TSH) 0.3-3.0 mIU/L
* Patient is scheduled or being considered for surgical resection of the nodule
* I-123 planar and Single Photon Emission Computed Tomography (SPECT)/Computed Tomography (CT) can be scheduled at least 2 days after biopsy and before surgery

Exclusion Criteria:

* Recent iodinated contrast, including intravenous (IV) and oral CT contrast or interventional vascular or cardiac study (within 6 weeks)
* Hurthle cell adenoma
* Current thyroid hormone supplementation
* Current use of anti-thyroid medications (methimazole or propylthiouracyl)
* Less than 2 days after thyroid nodule FNA/biopsy
* Presence of another nodule of similar size in the same area of thyroid lobe, which could impair localization of the nodule on SPECT/CT images
* Less than 2/3 of normal thyroid tissue present in either thyroid lobe without nodules
* Positive pregnancy test
* All women who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic patients with biopsy-proven indeterminate follicular thyroid lesions scheduled for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to study completion, up to one year
  Adverse events will be assessed while patients are in the nuclear medicine division undergoing positron emission tomography/computed tomography imaging.
Iodine-123 uptake | Up to study completion; up to one year
  We will compare the intensity of uptake in malignant versus benign lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta M. Durski, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials